CLINICAL TRIAL: NCT01003704
Title: Incidence of Phantom Limb Pain and Method of Anesthesia After Lower Extremity Amputation
Status: Completed | Type: Observational
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Chandramouli Iyer, MD, Veterans Affairs North Texas Health Care System
Other Study IDs: 09-059
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- General Anesthesia only
  Interventions: Procedure: Lower extremity amputation
- Peripheral nerve block
  Interventions: Procedure: Lower extremity amputation
- spinal
  Interventions: Procedure: Lower extremity amputation

INTERVENTIONS:
Procedure: Lower extremity amputation

SUMMARY:
Phantom limb pain (pain originating from where an amputated limb once was) is a common occurrence after lower extremity amputations, with some sources noting incidence to be as high as 60-80% six months after surgery. This pain can eventually subside, however, cases have been reported of incidence 10 years after surgery. This pain is not only physically detrimental, but can also be psychologically detrimental after a difficult to accept change in the body. Prior studies have been performed using regional anesthetic techniques (including spinals and epidurals) and different medications to attempt to reduce the incidence of phantom limb pain, however, the data have been mostly inconclusive. Of interest, prior studies have not addressed peripheral nerve blocks, a method of anesthesia/analgesia more commonly employed for amputations recently. The purpose of our retrospective study is to look at the incidence of phantom limb pain at our institution over a two year period to determine if peripheral nerve blocks result in a significantly reduced incidence compared to other techniques (spinal, epidural, general anesthesia only). In addition, there is little data on relation of reason for amputation and presence of preoperative neuropathy and incidence of phantom pain. As secondary endpoints, the investigators wish to investigate if certain reasons for amputation (trauma, peripheral vascular disease, diabetes, and others) and/or neuropathy lead to a higher incidence of phantom limb pain. The results of this study could impact future management of patients who are to receive amputations and may lead to further prospective studies on the topics involved.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive lower extremity amputation

Exclusion Criteria:

* Death or incapacitating medical condition since surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who receive lower extremity amputation
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs North Texas Health Care System, Dallas, Texas, United States